CLINICAL TRIAL: NCT03895801
Title: A Randomized, Double-blind, Double-dummy, Active-controlled, Multicenter, 2-part Phase II Study on Replacement of Steroids by IFX-1 in Active Granulomatosis With Polyangiitis (GPA) and Microscopic Polyangiitis (MPA)
Brief Title: Study of IFX-1 to Replace Steroids in Patients With Granulomatosis With Polyangiitis and Microscopic Polyangiitis.
Acronym: IXchange
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IFX-1-P2.5
Record Dates: First submitted 2019-03-08; First posted 2019-03-29 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Granulomatosis With Polyangiitis (GPA); Microscopic Polyangiitis (MPA)
Keywords: granulomatosis; polyangiitis; corticosteroid; replacement; glucocorticoid
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Systemic Vasculitis | interventions — vilobelimab; Glucocorticoids; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A Experimental + active comparator (Experimental): IFX-1 + reduced dose GC
  Interventions: Drug: IFX-1; Drug: Glucocorticoid (GC)
- Group B Placebo + active comparator (Active Comparator): Placebo-IFX-1 + standard dose GC
  Interventions: Drug: Placebo-IFX-1; Drug: Glucocorticoid (GC)
- Group C Experimental + placebo comparator (Placebo Comparator): IFX-1 + Placebo-GC
  Interventions: Drug: IFX-1; Drug: Placebo-Glucocorticoid (Placebo-GC)

INTERVENTIONS:
Drug: IFX-1 — intravenously administered
  Other Names: CaCP29
  Arms: Group A Experimental + active comparator; Group C Experimental + placebo comparator
Drug: Placebo-IFX-1 — intravenously administered
  Other Names: Placebo
  Arms: Group B Placebo + active comparator
Drug: Glucocorticoid (GC) — orally administered
  Other Names: Prednisone
  Arms: Group A Experimental + active comparator; Group B Placebo + active comparator
Drug: Placebo-Glucocorticoid (Placebo-GC) — orally administered
  Other Names: Placebo
  Arms: Group C Experimental + placebo comparator

SUMMARY:
The purpose of the study is to evaluate the efficacy of IFX-1 treatment as replacement for glucocorticoid (GC) therapy in subjects with polyangiitis (GPA) or microscopic polyangiitis (MPA).

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasmic antibody-associated vasculitis (AAV) is a group of potentially life-threatening autoimmune diseases. Preclinical data demonstrate that primed neutrophils are activated by anti-neutrophil cytoplasmic antibody (ANCA) and generate C5a that engages C5a receptors on neutrophils. Patients with ANCA-related disease have elevated plasma and urine levels of C5a in active disease but not in remission. IFX-1 is as a monoclonal antibody specifically binding to the soluble human complement split product C5a, which results in nearly complete blockade of C5a induced biological effects. Therefore, IFX-1 may be effective in the treatment of subjects with AAV.

In this Phase II study of 20 to 55 subjects with granulomatosis with GPA and MPA, IFX-1 will be administered in combination with reduced dose glucocorticoids or a placebo glucocorticoid compared with standard dose glucocorticoids.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA)
* Have ≥ 1 "major" item, or ≥ 3 other items, or ≥ 2 renal items on the Birmingham Vasculitis Activity Score Version 3 (BVASv3).
* Newly diagnosed or relapsed GPA or MPA that requires treatment with Cyclophosphamide (CYC) or Rituximab (RTX) plus GCs.
* Glomerular filtration rate ≥ 20 mL/min/1.73 m².

Exclusion Criteria:

* Any other multi-system autoimmune disease.
* Require mechanical ventilation at screening.
* Known hypersensitivity to any investigational medicinal product and/or any excipient.
* Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption.
* Have required management of infections, as follows (a) Chronic infection requiring anti-infective therapy within 3 months before screening. (b) Use of intravenous antibacterials, antivirals, anti-fungals, or anti-parasitic agents within 30 days of screening
* Current and/or history (within the previous 5 years) of drug and/or alcohol abuse and/or dependence.
* Evidence of Hep B, C and/ or HIV infection. Only subjects with documented negative historical results (within 4 weeks before screening) for Hep B,C Virus and HIV or a negative test by Screening can be included into the study.
* Abnormal laboratory findings at screening
* Current or history of malignancy, lymphoproliferative, or myeloproliferative disorder
* Received CYC or RTX within 12 weeks before screening or within 12 weeks before CYC or RTX is started for remission induction within 2 weeks before screening.
* Received > 3 g cumulative intravenous GCs within 4 weeks before screening.
* Received an oral daily dose of a GC of > 10 mg prednisone-equivalent for more than 6 weeks continuously prior to screening.
* Received an oral daily dose of a GC of > 80 mg prednisone equivalent within 2 weeks before screening.
* Received a CD20 inhibitor, anti-tumor necrosis factor treatment, abatacept, alemtuzumab, any other experimental or biological therapy, intravenous immunoglobulin (Ig) or plasma exchange, antithymocyte globulin, or required renal dialysis within 12 weeks before screening.
* Received a live vaccination within 4 weeks before screening
* Either active or latent tuberculosis treatment is ongoing.
* Pregnant or lactating.
* Abnormal electrocardiogram.
* Female subjects of childbearing potential unwilling or unable to use a highly effective method of contraception
* Participation in an investigational clinical study during the 12 weeks before screening.
* Male subjects with female partners of childbearing potential unwilling to use contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anja Pfaff, PhD, Study Director — InflaRx GmbH; Peter A. Merkel, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (66):
- Belgium (2):
  - Clinical Site, Leuven
  - Clinical Site, Liège
- Czechia (2):
  - Clinical Site, Hradec Králové
  - Clinical Site, Prague
- France (9):
  - Clinical Site, Angers
  - Clinical Site, Brest
  - Clinical Site, Créteil
  - Clinical Site, Grenoble
  - Clinical Site, Lille
  - Clinical Site, Montpellier
  - Clinical Site, Paris
  - Clinical Site, Pessac
  - Clinical Site, Poitiers
- Germany (14):
  - Clinical Site, Jena, Thuringia
  - Clinical Site, Aachen
  - Clinical Site, Berlin
  - Clinical Site, Cologne
  - Clinical Site, Dresden
  - Clinical Site, Essen
  - Clinical Site, Freiburg im Breisgau
  - Clinical Site, Hanover
  - Clinical Site, Kirchheim unter Teck
  - Clinical Site, Leipzig
  - Clinical Site, Ludwigshafen
  - Clinical Site, Mannheim
  - Clinical Site, Münster
  - Clinical Site, Stuttgart
- Italy (8):
  - Clinical Site, Catania
  - Clinical Site, Lecco
  - Clinical Site, Messina
  - Clinical Site, Milan
  - Clinical Site, Monza
  - Clinical Site, Pavia
  - Clinical Site, Pisa
  - Clinical Site, Verona
- Netherlands (2):
  - Clinical Site, Maastricht
  - Clinical Site, Rotterdam
- Russia (8):
  - Clinical Site, Kemerovo
  - Clinical Site, Moscow
  - Clinical site, Moscow
  - Clinical Site, Orenburg
  - Clinical Site, Petrozavodsk
  - Clinical site, Saratov
  - Clinical Site, Saratov
  - Clinical Site, Yaroslavl
- Spain (7):
  - Clinical Site, Alcorcón
  - Clinical Site, Badalona
  - Clinical Site, Barcelona
  - Clinical site, Barcelona
  - Clinical Site, Fuenlabrada
  - Clinical Site, L'Hospitalet de Llobregat
  - Clinical Site, Seville
- Sweden (3):
  - Clinical Site, Gothenburg
  - Clinical Site, Stockholm
  - Clinical Site, Uppsala
- Switzerland (2):
  - Clinical Site, Sankt Gallen
  - Clinical Site, Zurich
- United Kingdom (9):
  - Clinical Site, Aberdeen
  - Clinical Site, Cambridge
  - Clinical Site, Cardiff
  - Clinical Site, Leicester
  - Clinical Site, London
  - Clinical Site, Portsmouth
  - Clinical Site, Preston
  - Clinical Site, Reading
  - Clinical Site, Sheffield

RESULTS

PARTICIPANT FLOW:
Groups:
- IFX-1 + Placebo-GC: IFX-1: 800 mg intravenously administered on Days 1, 4, and 8, and then every other week from Week 2 (Day 15) to Week 16; Placebo-Glucocorticoid (Placebo-GC): orally administered daily
- Placebo-IFX-1 + Standard Dose GC: Placebo-IFX-1: Placebo infusion intravenously administered on Days 1, 4, and 8, and then every other week from Week 2 (Day 15) to Week 16; Glucocorticoid (GC): starting dose of 60 mg daily orally administered, then tapered down
- IFX-1 + Reduced Dose GC: IFX-1: 800 mg intravenously administered on Days 1, 4, and 8, and then every other week from Week 2 (Day 15) to Week 16; Glucocorticoid (GC): starting dose of 30 mg daily orally administered, then tapered down
Period: Overall Study
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Started | 18 | 24 | 15
Completed | 16 | 22 | 13
Not Completed | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- IFX-1 + Placebo-GC: IFX-1: intravenously administered; Placebo-Glucocorticoid (Placebo-GC): orally administered
- Placebo-IFX-1 + Standard Dose GC: Placebo-IFX-1: intravenously administered; Glucocorticoid (GC): orally administered
- IFX-1 + Reduced Dose GC: IFX-1: intravenously administered; Glucocorticoid (GC): orally administered
- Total: Total of all reporting groups
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC | Total
Number analyzed (Participants) | 18 | 24 | 15 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (11.4) | 55.0 (12.3) | 58.5 (14.0) | 57.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 5 | 17
  Male | 12 | 18 | 10 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 17 | 24 | 15 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 18 | 24 | 15 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
AAV disease type [Count of Participants; unit: Participants] — AAV = anti-neutrophil cytoplasmic antibody-associated vasculitis
  Participants
    Granulomatosis with polyangiitis (GPA) | 10 | 16 | 11 | 37
    Microscopic polyangiitis (MPA) | 8 | 8 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Clinical Response
Description: Efficacy Endpoint: Percentage of subjects achieving clinical response (reduction in Birmingham Vasculitis Activity Score version 3 [BVASv3] of ≥50% compared to baseline and no worsening in any body system). Subjects who received rescue therapy after Day 1 or discontinued due to related adverse event, lack of efficacy or progressive disease are considered as non-responders at all subsequent visits. The BVASv3 score ranges from 0 to 63 with higher values representing higher disease activity.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 18 | 23 | 13
Participants | 16 | 22 | 10

2. Secondary Outcome: Percentage of Subjects With Clinical Remission
Description: Efficacy endpoint: Percentage of subjects with clinical remission, defined as having a BVASv3 = 0. Subjects who received rescue therapy after Day 1 or discontinued due to related adverse event, lack of efficacy or progressive disease are considered as non-responders at all subsequent visits. The BVASv3 score ranges from 0 to 63 with higher values representing higher disease activity.
Time Frame: Week 16
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 18 | 23 | 13
Participants | 14 | 20 | 10

3. Secondary Outcome: Change From Baseline in BVASv3 Total Score
Description: Efficacy endpoint: Absolute Change from baseline (= screening assessment) in Birmingham Vasculitis Activity Score version 3 (BVASv3) total score; The BVASv3 score ranges from 0 to 63 with higher values representing higher disease activity. The total score is derived by summing up item scores according to the scoring manual for the BVASv3.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 16 | 22 | 12
score on a scale | -13.8 (4.1) | -14.7 (5.9) | -16.6 (5.8)

4. Secondary Outcome: Vasculitis Damage Index (VDI)
Description: Efficacy endpoint: Absolute values of VDI; The VDI total score ranges from 0 to 64 with higher scores indicating more organ damage since the onset of vasculitis. The total score is the number of present damage items.
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 16 | 22 | 12
score on a scale | 1.0 (1.0) | 1.5 (1.1) | 1.9 (1.8)

5. Secondary Outcome: Physician Global Assessment (PGA)
Description: Efficacy endpoint: Absolute values in PGA; Physician global assessment scale: 0 = Remission to 10 = Maximum activity;
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 16 | 22 | 12
score on a scale | 0.4 (1.0) | 0.1 (0.5) | 0.7 (1.8)

6. Secondary Outcome: Estimated Glomerular Filtration Rate
Description: Efficacy endpoint: Absolute values of estimated glomerular filtration rate (eGFR) in mL/min/1.73 m²; The eGFR was calculated by the central laboratory according to the Modified Diet in Renal Disease equation:
  eGFR = 175 x (serum creatinine, mg/dL)-1.154 x (age, years)-0.203 x (0.742 if female) x (1.212 if black)
Time Frame: Week 16
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 16 | 22 | 12
mL/min/1.73 m² | 50.2 (17.7) | 57.0 (22.8) | 51.2 (26.2)

7. Secondary Outcome: Number and Percentage of Subjects Who Had a Treatment-emergent Adverse Event (TEAE)
Description: Safety endpoint: Number and percentage of subjects who had a treatment-emergent adverse event (TEAE)
Time Frame: Week 24
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 18 | 24 | 15
Participants | 16 | 24 | 15

8. Secondary Outcome: Glucocorticoid Toxicity Index (GTI)
Description: Safety endpoint: The GTI total score ranges from -35 to 410 (because the bone domain is excluded in this study) with higher score indicating greater Glucocorticoid toxicity. Scoring was performed in the electronic case report form according to the corresponding scoring manual in "Development of a Glucocorticoid Toxicity Index (GTI) using multicriteria decision analysis." by Miloslavsky EM, Naden RP, Bijlsma JW, Brogan PA, Brown ES, Brunetta P, et al.
Time Frame: Week 16
Population: Safety Analysis Set (Data missing from 2 patients in IFX-1 + Placebo-GC group, from 2 patients in Placebo-IFX-1 + standard dose GC group, and from 3 patients in IFX-1 + reduced dose GC group)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 16 | 22 | 12
score on a scale | 0.8 (9.0) | 44.9 (41.5) | 26.1 (39.2)

9. Secondary Outcome: IFX-1 Plasma Concentrations (Pre-dose)
Description: Pharmacokinetics endpoint: IFX-1 plasma concentrations assessed prior to study drug administration at corresponding visit.
Time Frame: Week 16 (pre-dose)
Population: Safety Analysis Set (Data missing from 5 patients in IFX-1 + Placebo-GC group, from 7 patients in Placebo-IFX-1 + standard dose GC group, and from 7 patients in IFX-1 + reduced dose GC group)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 13 | 17 | 8
ng/mL | 67077.19 (77.33) | 47.80 (152.42) | 52597.85 (118.15)

10. Secondary Outcome: Plasma Concentrations of C5a
Description: Pharmacodynamics endpoint: Plasma concentrations of C5a
Time Frame: Week 16
Population: Full Analysis Set (Data missing from 4 patients in IFX-1 + Placebo-GC group, from 10 patients in Placebo-IFX-1 + standard dose GC group, and from 8 patients in IFX-1 + reduced dose GC group)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 14 | 14 | 7
ng/mL | 10.6816 (5.8505) | 39.2822 (25.6249) | 13.6320 (12.3040)

11. Secondary Outcome: IFX-1 Blocking Activity 10 nM
Description: Pharmacodynamics endpoint: IFX-1 blocking activity 10 nM
Time Frame: Week 16
Population: Full Analysis Set (Data missing from 4 patients in IFX-1 + Placebo-GC group, and from 7 patients in IFX-1 + reduced dose GC group, IFX-1 blocking activity was not assessed for patients in Placebo-IFX-1 + standard dose GC group)
Measure: Mean (Standard Deviation); unit: percentage of IFX-1 blocking activity
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 14 | 0 | 8
percentage of IFX-1 blocking activity | 100.571 (2.651) |  | 100.508 (10.051)

12. Secondary Outcome: IFX-1 Blocking Activity 2.5 nM
Description: Pharmacodynamics endpoint: IFX-1 blocking activity 2.5 nM
Time Frame: Week 16
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percentage of IFX-1 blocking activity
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
Number analyzed (Participants) | 14 | 0 | 8
percentage of IFX-1 blocking activity | 98.260 (16.731) |  | 121.881 (59.979)

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- IFX-1 + Placebo-GC: IFX-1: intravenously administered Placebo-Glucocorticoid (Placebo-GC): orally administered
- Placebo-IFX-1 + Standard Dose GC: Placebo-IFX-1: intravenously administered Glucocorticoid (GC): orally administered
- IFX-1 + Reduced Dose GC: IFX-1: intravenously administered Glucocorticoid (GC): orally administered
Arm/Group | IFX-1 + Placebo-GC | Placebo-IFX-1 + Standard Dose GC | IFX-1 + Reduced Dose GC
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/24 | 0/15
Serious Adverse Events (participants affected / at risk) | 5/18 | 4/24 | 3/15
Other Adverse Events (participants affected / at risk) | 15/18 | 23/24 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX-1 + Placebo-GC (N=18) | Placebo-IFX-1 + Standard Dose GC (N=24) | IFX-1 + Reduced Dose GC (N=15)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IFX-1 + Placebo-GC (N=18) | Placebo-IFX-1 + Standard Dose GC (N=24) | IFX-1 + Reduced Dose GC (N=15)
Nasopharyngitis (Infections and infestations) | 1 (1) | 6 (7) | 5 (6)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pustule (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 4 (4) | 2 (2)
Fat tissue increased (General disorders) | 1 (1) | 4 (5) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Condition aggravated (General disorders) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingivitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 6 (7) | 2 (2)
Haematoma (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Cyanosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Granulomatosis with polyangiitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
White coat hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (5) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Mood swings (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased interest (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heavy exposure to ultraviolet light (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Corneal erosion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dacryoadenitis acquired (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Secondary immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT03895801/Prot_SAP_000.pdf